CLINICAL TRIAL: NCT05225441
Title: National Investigation in College and High School Among Adolescents on Health and Substances at the FSEF
Acronym: EnCLASS-FSEF
Status: Completed | Type: Observational
Sponsor: Fondation Santé des Étudiants de France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02640-41
Record Dates: First submitted 2022-01-17; First posted 2022-02-04 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2021-12

CONDITIONS: Psychiatric Disorder; Somatic Symptom; Traumatic Injury
Keywords: clinical epidemiology; Substance use and abuse; Psychiatric symptoms; Social disabilities; Health literacy
MeSH Terms: conditions — Mental Disorders; Medically Unexplained Symptoms; Wounds and Injuries; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
For the clinical component:

Describe the young people hospitalised in residential care at the FSEF, in particular through vulnerability factors and their psychosocial repercussions (school level, repetition, intensity of symptoms, irritability, nervousness, substance use (cannabis, alcohol, tobacco), social relationships, family relationships, well-being, level of health literacy, learning disorders)) and to compare them with young people from the general school population.

For the epidemiological aspect:

To study the construct validity of the EnCLASS questions aiming to characterize handicap situations in the general school population in both a population in situation of psychic handicap and of somatic handicap.

DETAILED DESCRIPTION:
Residential care in psychiatry in France, although recommended by the HAS and widely implemented, have been little evaluated In France, the residential care of the FSEF called "soins-études" have long been recognized as contributors to psychosocial rehabilitation. They hospitalize young people with mental and physical disabilities. They allow the continuation of hospital care associated with the resumption of schooling and the implementation of a training project integrated into the individualized care plan. Each year, around 1 500 young people are admitted to full-time hospitalization for "soins-études" in psychiatry or medicine (follow-up care and rehabilitation) within the FSEF. They benefit from comprehensive care, adapted to their needs, including care, maintenance or resumption of schooling and social reintegration in a peer group. A recent review of the literature showed that the provision of "soins-études" in psychiatry allows clinical improvement in nearly two-thirds of between more than 5 years after admissionit, and the resumption of schooling and a training project. The young people admitted at the FSEF generally have been receiving care for more than 3 years for chronic psychiatric disorders. Despite frequent school delays or periods of dropping out of school, a large majority of them had a school activity during the care.

However, it appears from this review that the characteristics of the young people received have never been compared with those of students in a traditional education course. Characterizing this population meets a need, as well as a strong institutional demand (FSEF, funders and national education).

The EnCLASS-FSEF survey will be rolled out with the national EnCLASS methodology in all the annexes of the National Education schools integrated into the 13 FSEF care-study clinics (therefore on the total population in care-studies of the FSEF educated in secondary school) - making it possible to describe and compare the patients treated in care studies with the general school population.

ELIGIBILITY:
Inclusion Criteria:

* Student cared for in college and high school studies in the 13 clinics of the FSEF,
* From 11 years old,
* Non-opposition of the student to his participation in the study and to the use of his data (and of their parents for minor students).

Exclusion Criteria:

* Student opposition to participating in the study (or their parents for underage students).

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All young people hospitalized in care-study in the 13 clinics in the FSEF (i.e. around 1,500) over the period from March to June 2022.
Sampling Method: Non-Probability Sample
Enrollment: 598 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
description of the study population | inclusion
  Describe the young people taken into "soins étude" at the FSEF for a psychiatric pathology or for a somatic pathology, in particular through characteristic vulnerability factors and their psychosocial repercussions (school level, repetition, intensity of symptoms, irritability, nervousness, consumption of toxicants (cannabis, alcohol, tobacco), ease of having friends, quality of family relationships, well-being, level of health literacy, "dys" disorders)) and comparison with young people from the general school population. This description and comparison will be carried out thanks to the answers of the young people to the questionnaire of the national survey (identical questionnaire for the population of the FSEF and the national population).

SECONDARY OUTCOMES:
comparison | inclusion
  Compare the levels of psychological symtoms the FSEF population to the general population (response of young people to specific questions on the subject in the national survey questionnaire).
frequency | inclusion
  Frequency of various psychiatric disorders within the FSEF population and description of psychotropic treatments received. Data will be collected both through young people's responses to specific questions aimed at the FSEF population and both from the participants' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Godart, Study Director — Fondation Santé des Etudiants de France
Locations (1):
- Godart Nathalie, Paris, France

IPD SHARING:
Plan to Share IPD: No